CLINICAL TRIAL: NCT01251328
Title: Near Infrared Spectroscopy in Aortic Valve Replacement
Acronym: INSERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Principal Investigator, N Patrick Mayr, MD, Deutsches Herzzentrum Muenchen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE DHM-AN-OR-2010/01
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Aortic Valve Stenosis; Transcatheter Aortic Valve Implantation; Eligibility for Both Anaesthetic Methods
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- General anaesthesia (Active Comparator): General anaesthesia is performed under standardized conditions
  Interventions: Procedure: General anaesthesia
- Sedation (Active Comparator): Sedation is performed under standardized conditions
  Interventions: Procedure: Sedation

INTERVENTIONS:
Procedure: General anaesthesia — general anaesthesia is performed according to the hospitals standard
  Arms: General anaesthesia
Procedure: Sedation — Sedation is performed according to the hospitals standard
  Arms: Sedation

SUMMARY:
Transcatheter aortic valve implantation (TAVI) is an alternative for patients, that are considered to be too sick for conventional aortic valve replacement. There is no conclusive opinion about the best anesthesiologic management of these patients. Sedation and general anaesthesia are both adequate and the current literature shows no benefit towards one of these methods.

This study wants to investigate the influence of these two anesthesiologic managements on the cerebral oxygen saturation during the "rapid pacing"-period during valvuloplasty. The patients are randomised allocated to one of these two anaesthesiological managements. The investigators use the Near-Infrared Spectroscopy (NIRS) to measure the cerebral oxygen saturation. Parallel there will be a measurement of cerebral biomarkers to monitor cerebral hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* transcatheter aortic valve implantation

Exclusion Criteria:

* denial by patient
* denial by screening anaesthesist
* active neurodegenerative disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygen desaturation during the "rapid pacing" period and periprocedural | up to 48 hours
  Biomarkers for cerebral ischemia will be measured up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Patrick N Mayr, MD, Principal Investigator — Deutsches Herzzentrum München, Department of Anaesthesiology, Technische Universität München
Locations (1):
- Deutsches Herzzentrum München, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Mayr NP, Hapfelmeier A, Martin K, Kurz A, van der Starre P, Babik B, Mazzitelli D, Lange R, Wiesner G, Tassani-Prell P. Comparison of sedation and general anaesthesia for transcatheter aortic valve implantation on cerebral oxygen saturation and neurocognitive outcomedagger. Br J Anaesth. 2016 Jan;116(1):90-9. doi: 10.1093/bja/aev294. Epub 2015 Sep 29. PMID 26424178